CLINICAL TRIAL: NCT05697328
Title: Pseudoephedrine Prophylaxis for Prevention of Middle Ear Barotrauma in Hyperbaric Oxygen Therapy
Brief Title: Barotrauma in Hyperbaric Oxygen Therapy
Acronym: HBOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John Muir Health (Other)
Responsible Party: Principal Investigator, Jacinta Showers, Principal Investigator, John Muir Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22-10-01
Record Dates: First submitted 2022-12-26; First posted 2023-01-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Barotrauma
Keywords: hyperbaric oxygen therapy
MeSH Terms: conditions — Barotrauma | interventions — Pseudoephedrine

STUDY DESIGN:
Intervention Model Description: prospective randomized double-blind placebo control study design (enrollment ratio 1:1)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind placebo control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pseudoephedrine (Experimental): over the counter pseudoephedrine
  Interventions: Drug: Pseudoephedrine Pill
- Placebo (Placebo Comparator): pharmacy created placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pseudoephedrine Pill — One-time 60mg dose given orally between 45-120 minutes prior to hyperbaric oxygen therapy
  Other Names: Sudafed
  Arms: Pseudoephedrine
Drug: Placebo — One time dose given orally between 45-120 minutes prior to hyperbaric oxygen therapy
  Arms: Placebo

SUMMARY:
The purpose of this research is to study whether the use of pseudoephedrine can help prevent middle ear trauma during HBOT. Pseudoephedrine is an approved drug that is used for temporary relief of nasal or sinus pain and pressure.

DETAILED DESCRIPTION:
Subjects will be asked to take a pill (pseudoephedrine or placebo) between 45 and 120 minutes before hyperbaric oxygen therapy. Subjects' ears will be examined before and after therapy and be asked to assess ear pain. There will be no further tests or procedures after completion of therapy session and ear examinations.

ELIGIBILITY:
Inclusion Criteria:

* New patient requiring HBOT (either inpatient or outpatient)
* Age greater than or equal to 18 years and less than 80 years
* Fluent in English
* Full decision capacity
* Able and medically cleared to swallow a pill

Exclusion Criteria:

* Enrollment would delay hyperbaric therapy more than 30 minutes in patients with emergent indications (example: Central Retinal Arterial Occlusion, Carbon Monoxide, Air Gas Embolism)
* Contraindication to pseudoephedrine (monoamine oxidase inhibitors (MAOI) use, pregnancy, glaucoma, heart disease, allergy to drug class)
* Systolic Blood Pressure >160
* Diastolic Blood Pressure > 90
* Heart Rate >100
* Decongestant/antihistamine/pseudoephedrine/nasal steroid/oxymetazoline use within 12 hours.
* Prisoner
* Intubated
* Unable to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Compare changes in self-reported ear pain during hyperbaric oxygen therapy | 45-60 minutes
  Patients to describe pain on a numerical scale before, during and after hyperbaric oxygen therapy

SECONDARY OUTCOMES:
Incidence of completed compression | 1 minute
  Compare frequency of complete versus aborted hyperbaric oxygen therapy session due to pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jacinta Showers, RN, Principal Investigator — John Muir Health
Locations (1):
- John Muir Health, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No